CLINICAL TRIAL: NCT07307885
Title: The Effect of Photobiomodulation on Pressure Ulcers: A Randomized Controlled Trial
Brief Title: The Effect of Photobiomodulation on Pressure Ulcers
Acronym: Pressure Ulcer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Collaborators: Fenerbahce University (Other); Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hülya Elmalı Şimşek, Asst Prof, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ankaramedipol; university (Registry Identifier: Ankara Medipol University)
Record Dates: First submitted 2025-12-08; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pressure Ulcer (PU)
Keywords: photobiomodulation; Pressure Ulcer; wound care
MeSH Terms: conditions — Pressure Ulcer | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photobiomodulation group (Experimental): photobiomodulation intervention group
  Interventions: Device: photobiomodulation
- control group (No Intervention): routine hospital care

INTERVENTIONS:
Device: photobiomodulation — The effectiveness of photobiomodulation application in chronic wound healing will be evaluated.
  Arms: photobiomodulation group

SUMMARY:
Photobiomodulation Group (Intervention Group):

Before the intervention, the patient's skin sensitivity to light will be tested by applying light for 3 minutes to one-fourth of the forearm skin. If redness occurs and persists for more than 2 hours, this indicates photosensitivity, and the intervention will not be performed.

The Patient Information Form will be completed during the first meeting with the patients included in the study. Subsequently, blood values will be determined, the Patient Assessment Form will be filled out, vital signs will be measured, and then the intervention will begin. After routine wound care/cleaning procedures in the intensive care unit, without applying any medication, cream, or lotion to the wound area, red light (660 nm wavelength) will be applied to the wound area for 5 minutes at a distance of 55 cm during the first 3 days, and for 10 minutes at the same distance on the following days. This application will continue once daily for 14 days. Wound assessments will be performed, and photographs will be taken on Day 1, Day 4, Day 7, and Day 14 (Baracho et al., 2021; Viecelli et al., 2024; Lima et al., 2020).

Control Group:

The Patient Information Form will be completed during the first meeting with the patients included in the study. Subsequently, blood values will be determined, the Patient Assessment Form will be filled out, and vital signs will be measured. No intervention will be performed other than the routine wound care procedure carried out in the intensive care unit. Wound assessments will be performed, and photographs will be taken on Day 1, Day 4, Day 7, and Day 14, in the same manner as in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage II pressure ulcers
* Patients without any skin disease
* Patients with albumin, platelet, and blood glucose levels within normal ranges
* Patients who will stay in the intensive care unit for 14 days or longer
* Patients with a BMI of 35 or below
* Patients with vital signs within normal limits
* Patients with an oxygen saturation level of 90% or above

Exclusion Criteria:

* Patients who do not consent to participate in the study
* Patients with severe nutritional problems and those who are cachectic
* Patients with severe edema (+4 or above)
* Patients with diabetes mellitus
* Patients who show photosensitivity in the light sensitivity test
* Patients with metastatic tumors, high fever, thromboangiitis obliterans, vascular insufficiency, active tuberculosis, acute soft tissue infection, pregnancy, bleeding tendency, skin sensory disorders, or skin allergies
* Patients with acute injuries within the past 72 hours
* Patients with a pacemaker, defibrillator, or other electronic implants
* Patients taking medications known to cause photosensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
The healing of pressure sores in the patients in the experimental group will be faster and more effective than in the control group. | 14 days
  This application will be continued once a day for 14 days and wound evaluation will be made and wound photographs will be taken on days 1, 4, 7 and 14. Wound assessment will be based on Pressure Ulcer Scale for Healing-PUSH and wound measurement(diameter).

IPD SHARING:
Plan to Share IPD: Undecided